CLINICAL TRIAL: NCT03447782
Title: Endogenous Modulation and Central Sensitization in New Daily Persistent Headache ( NDPH ) in Children
Acronym: EMCS-NDPH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alyssa Lebel, MD, Director, Chronic Headache Program, Boston Children's Hospital ( BCH ); Associate Professor of Anesthesiology, HMS, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P00026929
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: New Daily Persistent Headache (NDPH)
Keywords: New Daily Persistent Headache; Chronic Headache
MeSH Terms: conditions — Headache Disorders | interventions — Naltrexone; Dietary Fiber; Powders

STUDY DESIGN:
Intervention Model Description: This group includes patients reviewed after 3 months of observational study with NDPH who have not improved clinically-they will take naltrexone, 4.5 mg, for 3 months. The other group includes healthy control patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NDPH Persistent (Experimental): Patients will be evaluated in clinic 1 month after the phone call evaluation. At this time, patients will begin a 3 month trial of low-dose naltrexone (Naltrexone HCL powder compounded to provide 4.5mg once per day orally).
  Patients will be evaluated in clinic 3 months after beginning treatment with naltrexone.
  Interventions: Drug: Naltrexone HCl (Bulk) Powder
- Healthy Controls (No Intervention): These participants will be in the research study for the initial visit only. They will be evaluated by a physician or nurse practitioner

INTERVENTIONS:
Drug: Naltrexone HCl (Bulk) Powder — For the NDPH Persistent group, patient will take naltrexone, 4.5 mg, po 1 time/day for three months-Naltrexone will be compounded from Naltrexone HCL powder
  Arms: NDPH Persistent

SUMMARY:
New daily persistent headache (NDPH) is a primary headache disorder characterized by the daily and unremitting headache pain patients experience with a distinct onset. Despite the known significant impairment associated with NDPH, the process by which some patients with NDPH recover within months while others do not is unknown.

The investigators propose to refine the clinical definition and suggest a novel mechanism underlying new daily persistent headache (NDPH) in adolescents. They further aim to investigate low-dose naltrexone for the treatment of new daily persistent headache. Healthy controls will also be enrolled in order to investigate the existence of a biomarker for NDPH. Adolescents ages 10-17 will be recruited from Boston Children's Hospital Pediatric Headache Program.

DETAILED DESCRIPTION:
The purpose of this study is to investigate low-dose naltrexone for the treatment of new daily persistent headache (NDPH) in adolescents ages 10-17. New daily persistent headache (NDPH) is a primary headache disorder characterized by continuous pain experienced for at least 3 months from distinct onset. Patients with NDPH have compromised academic performance, school absence, anxiety, depressed mood, sleep impairment, family disruption, and high health care costs. Despite the known significant impairment associated with NDPH, the process by which some patients with NDPH recover within months while others do not is unknown. With the goal of enhancing the clinical definition of NDPH, investigators will describe differences between patients with NDPH and healthy controls.

Additionally, little is known about which medications effectively manage and treat NDPH. One proposed medication that may benefit children and adolescents with NDPH is low-dose naltrexone. Naltrexone is an anti-inflammatory agent, similar to the opioid antagonist naloxone. Naltrexone is an effective treatment for opioid addiction, however, it was recently discovered that when taken in low doses (1/10 of the typical dose) naltrexone is capable of reducing the severity of chronic pain symptoms. By acting on glial cells in the nervous system as well as other receptors in the brain, naltrexone is capable of exerting analgesic effects. With this analgesic property, it has been speculated that low-dose naltrexone may be an effective treatment for the management of several chronic pain conditions, including headache.

Although more research must be conducted to evaluate long-term effects of using low-dose naltrexone, prior studies show that there are little short-term consequences associated with using this drug as a form of treatment for chronic pain symptoms. Investigators aim to assess the efficacy and safety of low-dose naltrexone in the treatment of patients with NDPH.

ELIGIBILITY:
Inclusion Criteria:

1) Patients meeting clinical International Classification of Headache Disorders (ICHD-3 )classification for NDPH 2) Age 10-17 years, all sexes, races, and ethnicities 3) English speaking 4) Able to wean off headache prophylactic medication 2 weeks prior to start of Naltrexone trial (patient will still be able to use abortive medication throughout the duration of the study) 5) On stable psychotropic medication for mild anxiety and/or mood disturbance for 2 weeks

-

Exclusion Criteria:

1) Children and adolescents with significant chronic medical illness: Central Nervous systen (secondary headache disorder other than mild traumatic brain injury); Cardiac, Pulmonary other than stable asthma, Metabolic, Renal, Hepatic 2) Significant psychiatric disorder, such as major depression, somatization disorder, and psychosis 3) Pregnancy 4) Intellectual delay or cognitive limitations precluding completion of questionnaires or following instructions.

-

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa Lebel, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No healthy controls were able to be recruited as the COVID-19 pandemic caused the study to shut down.
Groups:
- NDPH Persistent: Patients will be evaluated in clinic 1 month after the phone call evaluation. At this time, patients will begin a 3 month trial of low-dose naltrexone (Naltrexone HCL powder compounded to provide 4.5mg once per day orally).
  Patients will be evaluated in clinic 3 months after beginning treatment with naltrexone.
  Naltrexone HCl (Bulk) Powder: For the NDPH Persistent group, patient will take naltrexone, 4.5 mg, po 1 time/day for three months-Naltrexone will be compounded from Naltrexone HCL powder
Period: Overall Study
Arm/Group | NDPH Persistent
Started | 45
Completed | 25
Not Completed | 20

BASELINE CHARACTERISTICS:
Population: The healthy control arm was not included here as COVID-19 necessitated the shut-down of this study and no healthy controls were able to be recruited.
Arm/Group | NDPH Persistent
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 36
  Other | 2
  Black or African American | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Native American or Alaskan Native | 0
  Unknown | 7
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: 1. A change in pain intensity scores and headache frequency from visit 1 (V1) compared to visit 4 (V4) for NDPH patients after naltrexone has been administered for approximately 3 months. The NRS (numerical rating scale) will be used, with a pain score between 0 to 10, with 0 being no pain and 10 being worst pain imaginable.
Time Frame: 3 months
Population: The healthy control arm was not included here because COVID-19 necessitated the shut-down of this protocol and no healthy controls were able to be recruited.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDPH Persistent
Number analyzed (Participants) | 25
score on a scale
  V1 Pain Rating | 5.82 (1.47)
  V4 Pain Rating | 4.92 (1.64)

2. Secondary Outcome: Functional Disability
Description: 1. A change in functional disability scores - The functional disability inventory (FDI) will be used to assess differences in disability pre- and post-naltrexone treatment for NDPH patients The FDI is a valid and reliable measure consisting of 15 items concerning perceptions of physical and psychosocial function. Total scores range from 0 to 60, with higher scores indicating greater disability.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDPH Persistent
Number analyzed (Participants) | 25
score on a scale
  FDI V1 | 15.16 (8.56)
  FDI V4 | 10.96 (8.46)

3. Secondary Outcome: Self- Perceived Pain Sensitivity
Description: A change in self-perceived pain sensitivity - The Pain Sensitivity Questionnaire (PSQ) will be used to assess differences in pain sensitivity pre- and post-naltrexone treatment, as well as between persistent patients and healthy controls. The Pain Sensitivity Questionnaire (PSQ) PSQ is a valid 17 item self-report measure of pain sensitivity. Each item is rated on a scale of 0 to 10, with 0 being no pain and 10 being worst pain imaginable. The PSQ will be used to assess differences in pain sensitivity pre- and post-naltrexone treatment, as well as between recovered and persistent patients.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NDPH Persistent
Number analyzed (Participants) | 25
units on a scale
  PSQ total V1 | 3.21 (1.03)
  PSQ total V4 | 3.22 (1.50)

ADVERSE EVENTS:
Time Frame: 4-7 months
Description: The healthy control arm was not included here because COVID-19 necessitated the shut-down of this protocol and no healthy controls were able to be recruited.
Arm/Group | NDPH Persistent
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
This trial had to shut down due to the emergence of the COVID-19 virus in 2020. Because of this, our sample size is smaller than anticipated and thus serves as a limitation of our trial. Additionally, healthy controls were extremely difficult to recruit for the study given the COVID-19 pandemic and thus we were unable to adequately compare NDPH patients to healthy controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT03447782/Prot_SAP_000.pdf